CLINICAL TRIAL: NCT06656429
Title: Outcome of Transforminal Epidural Injections in Patients with Lumbar Radicular Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mayo-1
Record Dates: First submitted 2024-10-18; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Lumbar Redicular Pain
MeSH Terms: interventions — Dexamethasone; Lidocaine; Solutions

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TFESI (Experimental): Lumbar Transforaminal Epidural Steroid Injections was administered, consisting of 4 mg dexamethasone and 0.33% lidocaine in a 3 ml solution.
  Interventions: Drug: Transforaminal Epidural Steroid Injections

INTERVENTIONS:
Drug: Transforaminal Epidural Steroid Injections — Transforaminal Epidural Steroid Injections
  Other Names: Lumbar transforaminal epidural steroid Injection was administered, consisting of 4 mg dexamethasone and 0.33% lidocaine in a 3 ml solution

SUMMARY:
Back pain is the most common chronic pain disorder of adult population. Lumbar radicular pain occurs due to irritation or compression of the nerve roots in the lower back. Various non-surgical methods can also be exercised that have been used to treat lumbar radicular pain since the ancient times. Despite the availability of various treatment options, achieving optimal pain relief and functional recovery remains challenging. Lumbar Transforaminal Epidural Steroid Injections (TFESI) are commonly used to manage this condition, but there is variability in patient response and limited data on the effectiveness of TFESI in different demographic and clinical subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Aged between 45 and 80 years
* Experiencing lumbar radicular pain

Exclusion Criteria:

* History of spinal fracture or previous spinal surgery
* Recurrent pain within 3 months of prior treatment
* Ongoing steroid therapy
* IKnown allergy to dexamethasone or lidocaine

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Pain score | 4-week
  Patients were monitored for four weeks post-treatment, with follow-up visits scheduled at 1 week and 4 weeks. Pain scores were reassessed using visual analog scale (scores between 1 to 10). Lower scores meant lower pain whereas higher scores meant higher degree of pain

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Zarak Awais, MBBS, Principal Investigator — Department of Orthopedic Surgery, Mayo Hospital, Lahore, Pakistan
Locations (1):
- Mayo Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No